CLINICAL TRIAL: NCT05191355
Title: Screening for Familial Hypercholesterolemia in Children Using the Blotter Method, or Dried Blood Spot
Brief Title: Screening for Hypercholesterolemia in Children Using Dried Blood Spot
Acronym: CHOLESPOT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0178; 2021-A02907-34 (Other: ID-RCB)
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia, Familial; Pediatrics
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects with familial hypercholesterolemia: blood test
  Interventions: Biological: blood test
- healthy subjects: blood test
  Interventions: Biological: blood test

INTERVENTIONS:
Biological: blood test — Blood spot collection for sampling

SUMMARY:
Purpose:

Heterozygous Familial Hypercholesterolemia (HeFH) is a common genetic disease responsible for premature atherosclerosis. Therefore, early diagnosis and initiation of a treatment early as at the age of eight years old are recommended to reduce cardiovascular risk. Child-parent screening based on plasma LDL-cholesterol has been proposed to identify patients with hypercholesterolemia. However, in children, venipuncture is often an obstacle for screening. This study aims to evaluate the performance and feasibility of a dried blood spot collection to screen hypercholesterolemia.

Method: The lipid profile of 30 healthy and 30 hypercholesterolemic patients will be determined using Dried Blood Spot (DBS) collection and veinipuncture.

The study is conducted in accordance with the principles of the Declaration of Helsinki. The children, their parents and patients will be informed about this study according to the French bioethics law and will be included only after their agreement

Hypothesis

* to evaluate the performance of the determination of total and LDL-cholesterol using a dried blood spot collection to screen hypercholesterolemia
* to evaluate the feasibility of a dried blood spot collection to screen hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* patients/kindreds in family with a documented history of hypercholesterolemia
* healthy subjects for controls

Exclusion Criteria:

* refusal to participate in the study
* For control patients: to have a known dyslipidemia

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with heterozygous familial hypercholesterolemia and healthy subjects
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of lipid profile (total cholesterol, LDL cholesterol concentrations) between venous blood and blotter method for sampling | Day 0
  study of the feasibility and accuracy of the blotter method to screen hypercholesterolemia

CONTACTS AND LOCATIONS:
Overall Officials: Noël PERETTI, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Dept of Endocrinology, Bron
  - Hospices Civils de Lyon, Service d'Hépatologie et de Gastro-Entérologie et Nutrition Pédiatrique, Bron